CLINICAL TRIAL: NCT07163650
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Center Study of Efsubaglutide Alfa in Patients Remaining Obese 6 Months After Metabolic Surgery
Brief Title: Evaluating Anti-Obesity Medications 6 Months After Metabolic Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-0631-01
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Weight Loss; Metabolic Surgery
Keywords: obesity; BMI; GLP-1 receptor agonist; Efsubaglutide Alfa; Metabolic surgery
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Pharmaceutical Preparations; Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Efsubaglutide Alfa group (Experimental): Receive guidance on diet and exercise throughout the program, started pharmacological intervention at enrollment for 24 weeks.
  Interventions: Drug: Efsubaglutide Alfa Injection; Behavioral: Diet and exercise guidelines
- control group (Sham Comparator): Receive guidance on diet and exercise throughout the program, without the use of drugs.
  Interventions: Behavioral: Diet and exercise guidelines

INTERVENTIONS:
Drug: Efsubaglutide Alfa Injection — Efsubaglutide Alfa was injected daily in the morning before meals Subcutaneous injection at a dose of 1 mg/week in the first two weeks, increased to 3 mg/week in week 3, increased to 6 mg/week in week 5, up to 9 mg/2 week in week 13.
  Other Names: Drug injection
  Arms: Efsubaglutide Alfa group
Behavioral: Diet and exercise guidelines — Participants followed a science-based diet and exercise program intervention.
  Other Names: Lifestyle guidelines

SUMMARY:
This clinical trial aims to evaluate the weight-loss efficacy and safety of efsubaglutide alfa in patients who remain obese 6 months after metabolic surgery.

DETAILED DESCRIPTION:
This study investigates the effects of efsubaglutide alfa intervention in patients with a body mass index (BMI) ≥28 kg/m² six months after metabolic surgery, aiming to determine whether it facilitates weight normalization and remission of obesity-related comorbidities, thereby assessing the weight-loss and metabolic benefits of early efsubaglutide alfa application in post-metabolic surgery obesity management.

ELIGIBILITY:
Inclusion Criteria:

* 6 months after metabolic surgery
* 18 years ≤ age ≤ 55 years
* Body Mass Index (BMI) ≥ 28 kg/m^2
* Voluntarily sign the informed consent form and agree to strictly adhere to the requirements and restrictions outlined in the informed consent form and this protocol throughout the entire study period.

Exclusion Criteria:

* Subjects suspected by the investigator of having a potential allergy to the study drug or its components, or those with a history of allergic constitution;

  * Use of any of the following drugs or treatments prior to screening:

    ● Glucagon-like peptide-1 (GLP-1R) agonists within 3 months prior to screening

    ● Use within 3 months prior to screening of any weight-affecting medications, including systemic corticosteroids, metformin, sodium-glucose cotransporter 2 (SGLT2) inhibitors, etc.;

    ● Use of weight-affecting herbal supplements, health products, or meal replacements within 3 months prior to screening;
    * Use of weight-loss medications within 3 months prior to screening or currently using such medications, e.g., sibutramine hydrochloride, orlistat, phentermine, etc.;
    * Participation in other clinical trials (receiving investigational drug treatment) within 3 months prior to screening.

      ③ History or evidence of any of the following conditions prior to screening:
    * History of depression; or history of severe psychiatric disorders such as schizophrenia, bipolar disorder, etc.;
    * Uncontrolled hypertension at screening despite at least 4 weeks of antihypertensive medication, defined as systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg;
    * History of malignancy at screening;
    * History of cardiac disease at screening: acute myocardial infarction, unstable angina, post-coronary artery bypass grafting, post-percutaneous coronary intervention, severe arrhythmia;
    * Hemorrhagic or ischemic stroke, or transient ischemic attack within 6 months prior to screening;
    * History or family history of medullary thyroid carcinoma, multiple endocrine neoplasia (MEN) type 2A or 2B at screening;
    * History of acute or chronic pancreatitis, or pancreatic injury at screening;
    * Presence of limb deformities or amputations preventing accurate measurement of height, weight, or other anthropometric parameters;
    * Major or moderate surgery, severe trauma, or severe infection within 1 month prior to screening, deemed unsuitable for study participation by the investigator;
    * History of suicidal tendencies or suicide attempts;
    * Anticipated surgery during the study period;
    * Participants testing positive for HIV antibodies, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, or syphilis antibodies at screening;
    * History of alcohol abuse within 1 month prior to screening, defined as average weekly alcohol intake exceeding 21 units for males or 14 units for females; ④ Presents clinically significant abnormalities on 12-lead electrocardiogram (ECG) at screening: - Second- or third-degree atrioventricular block - Long QT syndrome or QTcF > 450 ms - PR interval < 120 ms or PR interval > 220 ms - QRS > 120 ms QRS duration >120ms, left or right bundle branch block, Wolff-Parkinson-White syndrome, or other severe arrhythmias requiring treatment;

      * History of other risk factors for torsades de pointes, such as hypokalemia at screening, family history of long QT syndrome, or concomitant use of QT/QTc-prolonging medications at screening; ⑥ Blood donation volume and/or blood loss ≥400 mL within 3 months prior to screening, or hemoglobin <110 g/L (males) or <100 g/L (females); ⑦ Presence of any other factors deemed by the investigator to potentially affect the efficacy or safety evaluation of this study, rendering the subject unsuitable for participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in %TWL from baseline to endpoint | 24 weeks from enrollment
  %TWL = ([baseline weight - weight at follow-up]/baseline weight) × 100%. The measurement of body weight is in kilograms. %TWL represents the percentage of total weight loss, measured in percent. This indicator reflects the percentage of weight loss from the baseline. The mean and standard deviation of %TWL were calculated for subjects within each group. Subsequently, intergroup comparisons were performed to calculate p-values. If p < 0.05, pairwise comparisons were further conducted. Based on the final results, the differences in weight loss among groups were evaluated.

SECONDARY OUTCOMES:
Proportion of patients with different %TWL levels | 24 weeks from enrollment
  %TWL = ([baseline weight - weight at follow-up]/baseline weight) × 100%. The measurement of body weight is in kilograms. %TWL represents the percentage of total weight loss, measured in percent. This indicator reflects the proportion of patients achieving clinically meaningful %TWL thresholds (≥ 5%, ≥ 10%, ≥ 15%, and ≥ 20%). Then perform intergroup comparison to calculate the p-value and assess the weight loss difference between the two groups.
Proportion of patients with normal weight and overweight | 24 weeks from enrollment
  BMI = Weight / Height^2 Weight is measured in kilograms, height in meters, and BMI is expressed in kilograms per square meter. This indicator reflects percentage of patients with normal weight (BMI<24kg/m2) and overweight (BMI <28kg/m2) from baseline after intervention. Then perform intergroup comparison to calculate the p-value and assess the difference between the two groups.
Change in body composition from baseline to endpoint across patient groups | 24 weeks from enrollment
  Body composition (Including body fat, fat-free mass, skeletal muscle, etc.; in kilograms） Body composition values at the endpoint minus baseline values are used as the change metric to evaluate body composition changes (These indicators are used to assess the body composition improvement of patients) Complete data correction for each patient using baseline values, then calculate overall mean and SD by group. Subsequently perform intergroup comparisons to compute P-values; if P < 0.05, proceed with pairwise comparisons.
Remission Status of Obesity-Related Diseases | 24 weeks from enrollment
  Obesity-Related Diseases include: Diabetes Mellitus, Hypertension, Fatty Liver Disease, Hyperlipidemia and Hyperuricemia.
  Remission status was assessed based on the incidence of complications in patients at baseline and endpoint. Then perform intergroup comparison to calculate the p-value and assess the differences in disease remission between the two groups.
Changes in blood pressure from baseline to endpoint | 24 weeks from enrollment
  Difference between the endpoint blood pressure and the baseline value.(blood pressure in mmHg; This indicator is used to assess improvements in a patient's blood pressure.) Complete data correction for each patient using baseline values, then calculate overall mean and SD by group. Subsequently perform intergroup comparisons to compute P-values; if P < 0.05, proceed with pairwise comparisons.
Changes in fasting blood glucose from baseline to endpoint | 24 weeks from enrollment
  Difference between endpoint fasting blood glucose and baseline value (blood glucose in mmol/L; This indicator is used to assess improvements in patients' fasting blood glucose levels.) Complete data correction for each patient using baseline values, then calculate overall mean and SD by group. Subsequently perform intergroup comparisons to compute P-values; if P < 0.05, proceed with pairwise comparisons.
Change in HbA1c from baseline to endpoint across patient groups | 24 weeks from enrollment
  Difference between the endpoint HbA1c value and the baseline value (HbA1c in percentage, This indicator is used to assess improvements in a patient's HbA1c levels.) Complete data correction for each patient using baseline values, then calculate overall mean and SD by group. Subsequently perform intergroup comparisons to compute P-values; if P < 0.05, proceed with pairwise comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhuan W Feng, MD, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
No participant data are available